CLINICAL TRIAL: NCT07024901
Title: The Effectiveness of The Somatic Intervention 'Dance-Walk' on Body Awareness, Vitality, and Mental Health
Brief Title: The Effects of the Somatic Intervention 'Dance-Walk' on Body Awareness, Vitality, and Mental Health in Help-Seeking Adults: a RCT Study
Acronym: DANCEWALK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vilnius University (Other)
Responsible Party: Principal Investigator, Inga Truskauskaitė, Associate professor, Vilnius University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: (1.13 E) 250000-KT-33
Record Dates: First submitted 2025-06-09; First posted 2025-06-17 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Healthy; Psychological Distress; Stress; Depression Disorders; Anxiety; Well-being; Mental Health; Body Awareness; Vitality
Keywords: Mental Health; Depression; Anxiety; Stress; Psychological Distress; Emotional Well-being; Somatic Intervention; Body-Mind Intervention; Mind-Body Practice; Embodied Practice; Body Awareness; Interoception; Vitality; Subjective Vitality; Positive Mental Health; Well-being; Adults; Help-seeking Adults; Randomized Controlled Trial; RCT; Waitlist Control; Autonomic Nervous System; Emotion Regulation; Stress Reduction; Mindfulness; Self-Awareness
MeSH Terms: conditions — Anxiety Disorders; Psychological Well-Being; Depression; Emotional Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participated in the "Dance-Walk" intervention after baseline measurment
  Interventions: Behavioral: Dance-walk
- Waiting-list control (No Intervention): Participates in the "Dance-Walk" intervention after the last study measure

INTERVENTIONS:
Behavioral: Dance-walk — Dance-Walk is a 4-week somatic intervention combining movement, dance, and walking elements designed to enhance body awareness and emotional regulation. The program consists of 4 weekly group sessions, each lasting approximately 90-120 minutes. Sessions focus on helping participants connect with their body sensations through guided movement exercises that integrate dance movements with mindful walking practices. The intervention targets autonomic nervous system regulation and aims to improve interoceptive awareness, emotional expression, and stress management through embodied practices. Sessions are facilitated by trained practitioners and emphasize non-verbal emotional expression and somatic experiencing to promote mental health and vitality.
  Arms: Intervention group

SUMMARY:
The goal of this clinical trial is to learn if a movement program called "Dance-Walk" can improve body awareness, energy levels, and mental health in adults seeking mental health support. The main questions it aims to answer are:

Does Dance-Walk help people feel more connected to their bodies? Does Dance-Walk increase people's energy and vitality? Does Dance-Walk improve mental health by reducing depression, anxiety, and stress?

Researchers will compare people who do Dance-Walk right away to people who wait to do the program later to see if Dance-Walk works to improve mental health.

All participants will fill out online surveys about their mood, energy levels, and body awareness at the start of the study. Then, every participant will be randomly placed into one of two groups - one group will start Dance-Walk right away, the other will wait. Participants who will be assigned to the first group will attend 4 weekly Dance-Walk sessions that combine movement, dance, and walking. All participants will fill out the same surveys again after the 4-week program. Participants who will be assigned to the second group will get to do the Dance-Walk program after the first group finishes.

Each Dance-Walk session will focus on helping people tune into their body feelings and use movement to manage emotions and stress. The program is designed to help people feel more energetic and improve their overall mental well-being.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Seeking to improve emotional well-being or mental health
* Able to participate in light physical activity (walking and gentle movement)
* Able to read and understand Lithuanian language
* Willing to attend 4 weekly group sessions
* Able to complete online questionnaires
* Willing to be randomly assigned to either immediate intervention or waitlist group
* Able to provide informed consent

Exclusion Criteria:

* Under 18 years of age
* Current severe mental health crisis requiring immediate professional intervention
* Physical limitations that prevent participation in walking or gentle movement activities
* Unable to commit to attending 4 weekly sessions
* Currently participating in another research study involving mental health interventions
* Unable to access internet for completing online questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2025-03-12 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Multidimensional Assessment of Interoceptive Awareness Scale-2 (MAIA-2) (Mehling et al., 2018) | Baseline to immediately post-intervention (approximately 4 weeks)
  Assesses multiple dimensions of interoceptive awareness, including noticing (score range: 0-20), not-distracting (score range: 0-30), not-worrying (score range: 0-25), attention regulation (score range: 0-35), emotional awareness (score range: 0-25), self-regulation (score range: 0-20), body listening (score range: 0-15), and trusting (score range: 0-15). Higher scores indicate greater interoceptive awareness (better outcome).
Subjective Vitality Scale (SVS) (Ryan & Frederick, 1997) | Baseline to immediately post-intervention (approximately 4 weeks)
  Measures feelings of energy and aliveness (score range: 0-47). Higher scores indicate greater subjective vitality and energy levels (better outcome).

SECONDARY OUTCOMES:
Depression Anxiety Stress Scales-21 (DASS-21) (Lovibond & Lovibond, 1995) | Baseline to immediately post-intervention (approximately 4 weeks)
  Assesses symptoms of depression (score range: 0-21), anxiety (score range: 0-21), and stress (score range: 0-21). Higher scores indicate more mental health problems (worse outcome).
Positive Mental Health Scale (PMH-Scale) (Lukat et al., 2016) | Baseline to immediately post-intervention (approximately 4 weeks)
  Measures positive aspects of mental health, including emotional well-being, psychological well-being, and social well-being (score range: 0-27). Higher scores indicate better positive mental health (better outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Inga Truskauskaite, PhD, Principal Investigator — Vilnius University
Locations (1):
- Vilnius university, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lukat J, Margraf J, Lutz R, van der Veld WM, Becker ES. Psychometric properties of the Positive Mental Health Scale (PMH-scale). BMC Psychol. 2016 Feb 10;4:8. doi: 10.1186/s40359-016-0111-x. PMID 26865173
- [Background] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther. 1995 Mar;33(3):335-43. doi: 10.1016/0005-7967(94)00075-u. PMID 7726811
- [Background] Ryan RM, Frederick C. On energy, personality, and health: subjective vitality as a dynamic reflection of well-being. J Pers. 1997 Sep;65(3):529-65. doi: 10.1111/j.1467-6494.1997.tb00326.x. PMID 9327588
- [Background] Mehling WE, Acree M, Stewart A, Silas J, Jones A. The Multidimensional Assessment of Interoceptive Awareness, Version 2 (MAIA-2). PLoS One. 2018 Dec 4;13(12):e0208034. doi: 10.1371/journal.pone.0208034. eCollection 2018. PMID 30513087